CLINICAL TRIAL: NCT01462617
Title: A Single-centre. Double-blind, Placebo Controlled Three Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Single and Repeat Doses of Nebulised GSK2269557 in Healthy Male Subjects
Brief Title: Study to Investigate Safety, Tolerability, Pharmacokinetics & Pharmacodynamics of Single & Repeat Doses of GSK2269557
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 115117
Record Dates: First submitted 2011-10-06; First posted 2011-10-31 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Nemiralisib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pi3K (Experimental): Experimental
  Interventions: Drug: GSK2269557
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: GSK2269557 matching placebo

INTERVENTIONS:
Drug: GSK2269557 — Study Drug
  Arms: Pi3K
Drug: GSK2269557 matching placebo — Study Drug
  Arms: Placebo

SUMMARY:
The study will comprise three Parts:

Part A will consist of two cohorts of healthy male volunteers to assess the safety, tolerability and pharmacokinetics of ascending single doses of nebulised GSK2269557. Blinded safety and available PK data will be reviewed before each dose escalation.

Part B will be one cohort to examine the safety, tolerability and pharmacokinetics of a repeated dose of GSK2269557 given by nebuliser for 7 days in healthy male volunteers. The total daily dose will be the same as, or lower than, doses that are well tolerated in Part A.

Part C will consist of two cohorts of single nebulised doses in healthy male smokers, to assess pharmacodynamic endpoints in sputum and bronchoalveolar lavage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included at the Investigator's discretion provided the abnormality will not jeopardize subject safety or study integrity .
* Male between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until the follow up visit.
* Body weight greater than or equal to 55kg and BMI within the range 18-31 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcB < 450 msec
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin less than or equal to 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).

Additional inclusion criteria for healthy smokers Cohorts 4-5 (Part C)

* Subjects who are current smokers. Must have smoked in the 12-month period preceding the screening visit and have a pack history of greater than or equal to 5 pack years. [number of pack years = (number of cigarettes per day/20) x number of years smoked].
* Normal spirometry (FEV1 greater than or equal to 80% of predicted, FEV1/FVC ratio greater than or equal to 70%) at screening. Predictions should be according to ECCS equations

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A history of congestive heart failure, coronary insufficiency or cardiac arrhythmia or a finding on screening 24h Holter monitor that would contraindicate the subject's participation in the study.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

  • an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* The subject has received any type of vaccination within 3 weeks of their first dose of investigational product, or are expected to be vaccinated within 3 weeks after their last dose of investigational product.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy (including atopic asthma) that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Subjects who have asthma or a history of asthma.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2011-07-24 (Actual); Primary Completion 2012-03-26 (Actual); Study Completion 2012-03-26 (Actual)

PRIMARY OUTCOMES:
clinical monitoring of blood pressure and pulse rate | Day 1 until Day 8
clinical monitoring of cardiac parameters | Day 1 until Day 8
clinical monitoring of lung function | Day 1 until Day 8
clinical monitoring of safety laboratory data | Day 1 until Day 8
clinical monitoring of adverse events | Day 1 until Day 8

SECONDARY OUTCOMES:
Pharmacokinetics profile at predose, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 hours post-dose. Profile to include Cmas, Area Under the Curve, Tmax | Day 1 to Day 8
PD bimoarkers potentially to incldue PIP3, Akt, S6K, IFNy, IgE, CD62L and CD44. | Day 1 to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115117 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115117?search=study&search_terms=115117#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 115117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115117 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register